CLINICAL TRIAL: NCT00271089
Title: Collection of Hematopoietic Cells From Patients With Fanconi Anemia (FA) for Future Autologous Reinfusion and Research
Brief Title: Blood Cell Collection for Future Use in Individuals With Fanconi Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 378; CCHMCEH001; R01HL081499-01A1 (NIH)
Record Dates: First submitted 2005-12-29; First posted 2005-12-30 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2007-12

CONDITIONS: Fanconi Anemia
MeSH Terms: conditions — Fanconi Anemia

INTERVENTIONS:
Procedure: PBSC Collection
Procedure: Bone Marrow Harvest
Device: CliniMacs Cell Selection System

SUMMARY:
Fanconi anemia (FA) is a disease that affects an individual's bone marrow. It is caused by a defective gene in the CD34+ cells, which are responsible for producing various types of blood cells. Individuals with FA may experience fatigue, bleeding, and increased infections. The purpose of this study is to collect and purify blood cells from individuals with FA and store them for future therapeutic use.

DETAILED DESCRIPTION:
FA is a rare, inherited disease that is caused by a gene defect to the CD34+ cells. It primarily affects an individual's bone marrow, resulting in decreased production of blood cells. The lack of white blood cells affects an individual's ability to fight infections, the lack of platelets may result in bleeding, and the lack of red blood cells usually leads to anemia. FA is typically diagnosed in childhood, and there is a high fatality rate. This study will use two methods to collect, purify, and store participant's CD34+ cells for future use in case of severe bone marrow failure. The collected cells will also be used by researchers to better understand the causes of FA and to possibly develop new treatments.

This study will enroll individuals with FA. All participants will undergo a bone marrow biopsy within 3 months of study entry. Based on the results of this biopsy, participants will undergo either a bone marrow harvest procedure or a cytokine mobilized peripheral blood stem cell (PBSC) collection procedure. Prior to both procedures, medical history will be reviewed, blood will be drawn, liver and kidney function will be evaluated, and a physical examination will be performed. Participants who undergo the bone marrow harvest procedure will be admitted to the hospital, with a possible overnight stay for observation. The following day, participants will have a physical examination and blood draw for laboratory testing. A blood and/or platelet transfusion may be required following the procedure.

Participants who undergo the PBSC procedure will be required to receive injections of G-CSF, a protein found normally in the body, twice a day for 4 to 8 days prior to the procedure; G-CSF has been found to help increase the amount of CD34+ cells in the blood. Once the CD34+ level is within a certain range, the PBSC procedure will begin through an IV placed in the arm or a temporary collection catheter placed under the participants' collarbone. Blood cells will be collected, with some cells separated out and the remainder of the cells infused back into the participant. The length of this procedure will vary for each participant; it will take 3 to 6 hours a day, for 1 to 4 days. Participants may require blood and/or platelet transfusions prior to and during the procedure.

Following the bone marrow harvest and PBSC procedures, CD34+ cells will be isolated in a laboratory. The majority of the cells will be frozen and stored for future use by the participants. A small portion of the cells will be available for researchers to perform experimental research to better understand FA.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FA
* Normal bone marrow cytogenetics within 3 months of study entry
* Absolute neutrophil count (ANC) level greater than 750
* Hemoglobin level greater than 8 without transfusion
* Platelet level greater than 30,000 without transfusion
* Must weigh at least 7.5 kg

Exclusion Criteria:

* Myloid or lymphoid leukemia
* Cytogenic abnormalities
* HIV infected
* Neoplastic or non-neoplastic disease of any major organ system that would compromise the ability to withstand the collection procedure
* Uncontrolled infection
* Unable to tolerate general anesthesia
* Known adverse reaction to E. Coli
* Pregnant or breastfeeding

Ages: 1 Year to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-08; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
CD34+ cell collection

CONTACTS AND LOCATIONS:
Overall Officials: Stella Davies, MBBS, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Kelly PF, Radtke S, von Kalle C, Balcik B, Bohn K, Mueller R, Schuesler T, Haren M, Reeves L, Cancelas JA, Leemhuis T, Harris R, Auerbach AD, Smith FO, Davies SM, Williams DA. Stem cell collection and gene transfer in Fanconi anemia. Mol Ther. 2007 Jan;15(1):211-9. doi: 10.1038/sj.mt.6300033. PMID 17164793